CLINICAL TRIAL: NCT02545660
Title: The Use of QLF-D (Quantitative Light-induced Fluorescence-DigitalTM) as an Oral Hygiene Evaluation Tool to Assess Plaque Accumulation and Enamel Demineralisation in Orthodontics
Brief Title: The Use of Quantitative Light Induced Fluorescence Digital as an Oral Hygiene Evaluation Tool in Orthodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4984
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2015-09

CONDITIONS: Complication of Personal Oral Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLF Image (Experimental): At each of the three visits tooth brushing advice will be given. The participants in the QLF group will be shown the QLFD images.Standardized oral hygiene reinforcement shall be given based on the images. The oral hygiene instruction will focus on the areas of the teeth which require greater emphasis, as shown by the images. Thus the patients should benefit from this detailed instruction.
  Interventions: Other: QLF Image
- White light Image (Experimental): At each of the three visits tooth brushing advice will be given. The participants in the white light image group will be shown the White light images.Standardized oral hygiene reinforcement shall be given based on the White light images. The oral hygiene instruction will focus on the areas of the teeth which require greater emphasis, as shown by the images. Thus the patients should benefit from this detailed instruction.
  Interventions: Other: White Light Image

INTERVENTIONS:
Other: QLF Image — At each of the three visits tooth brushing advice will be given. The participants in the intervention group will be shown the QLFD images or white light images.Standardized oral hygiene reinforcement shall be given based on the images. The oral hygiene instruction will focus on the areas of the teeth which require greater emphasis, as shown by the images. Thus the patients should benefit from this detailed instruction.
  Arms: QLF Image
Other: White Light Image — At each of the three visits tooth brushing advice will be given. The participants in the white light image group will be shown white light images.Standardized oral hygiene reinforcement shall be given based on the images. The oral hygiene instruction will focus on the areas of the teeth which require greater emphasis, as shown by the images. Thus the patients should benefit from this detailed instruction.
  Arms: White light Image

SUMMARY:
During orthodontic treatment bacterial plaque readily accumulates on the teeth. This is because food easily accumulates around the braces and it is more difficult to clean when the braces are in place. The plaque accumulation can lead to demineralisation (white spots) developing on the teeth. This is the start of decay and can lead to permanent marks and fillings being required.Prior to the start of orthodontic treatment adequate oral hygiene is necessary.

During orthodontic treatment, it is important that patients have an excellent level of oral hygiene to prevent plaque accumulating and demineralisation occurring. However, adequate tooth brushing can be difficult to perform as the bacterial plaque is not easily visible. Thus patients may not be able to see which areas need better tooth brushing.

QLFD(Quantitative Light Induced Fluorescence Digital) is a noninvasive method that uses fluorescent light to illuminate the oral bacteria in plaque that are responsible for demineralisation. The purpose of this study is to use the QLFD camera to assess its ability to measure plaque accumulation and demineralisation before the start of orthodontic treatment. The study will also assess the QLFD camera as a tool to improve oral hygiene.

DETAILED DESCRIPTION:
Plaque is a contributing factor for the development of dental diseases including tooth decay and gum disease. Thus, an excellent standard of oral hygiene is required to ensure all plaque is removed from the teeth to reduce the risk of developing these diseases.

Plaque accumulation starts and is greatest at plaque stagnation sites, which tend to be at the gum margins. In orthodontic treatment, the brackets and archwires are significant plaque stagnation sites.Conventional tooth brushing is also more difficult compounding the increased plaque accumulation and retention.

It is very important that patients learn to recognize the presence of plaque to ensure optimal levels of oral hygiene are achieved. Frequently patients have difficulty localizing the deposits to enable optimal levels of oral hygiene.

Demineralisation occurs due to bacterial fermentation of dietary sugars, which produces acids. This leads to white marks developing on the tooth surfaces, which is the first stage of dental caries. The risk of demineralisation is increased during orthodontic treatment, as there tends to be greater plaque accumulation. Previous studies have reported prevalence rates of demineralisation during orthodontic treatment to be as high as 96%. The most visible front surfaces of the teeth are often the most severely affected which can have a detrimental impact on their appearance.

Early demineralisation can be reversible if plaque control is improved, however progresses cavities may develop which require restoration. The main form of management of demineralisation is prevention. This is mainly by having an excellent level of oral hygiene and having a diet with a limited number of sugar intakes.

During orthodontics, patients frequently find it difficult to detect the plaque around the braces, thus oral hygiene is often not adequate. This leads to greater plaque accumulation and an increased risk of developing demineralisation.

The QLFD Biluminator is a noninvasive novel device, based on previous QLF technology. In vitro and in vivo studies of the former QLF device demonstrated it to be appropriate for identifying demineralisation and longitudinal monitoring of mineral changes during orthodontics. The advantage of the new QLFD device is that it takes a white light image in addition to a QLF image. Having two images, taken nearly simultaneously, allows comparisons to be made and ensures consistency with regards to magnification and angulation. From these images, plaque accumulation and demineralisation can be measured. In addition, demineralisation can be detected on QLF images before it is evident on white light images, which is of great benefit to clinicians in detecting at risk patients.

This study aims to assess plaque accumulation and demineralisation using the new QLFD device before the start of orthodontic treatment. It will also assess its use as an oral hygiene evaluation tool to improve patients tooth brushing who have inadequate oral hygiene to start orthodontic treatment. White light and QLF images will be taken with the QLFD device and patients will be given focused oral hygiene advice based on these images.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will consent.
2. All participants will be in good health.
3. At least 11 years of age.
4. Patients with poor level of oral hygiene undergoing pre-treatment visits with the hygienist or a dentist.

Exclusion Criteria:

1. Patients with significant disabilities that may affect manual dexterity and oral hygiene practice.
2. Patients who have had antibiotics in the last two months.
3. Patients with full coronal coverage restorations.
4. Patients with visually cavitated lesions.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
To find difference in plaque accumulation (ΔR30)between the White light group and QLF groups. | 6 Months
  The difference in plaque accumulation (ΔR30) between the White light group and QLF groups from visit 1 to visit 3 will be measured. QLFD camera will take QLF(blue light) and WL (white light) photographs. Either white light image or QLF image (based on which group patient is randomized to) will be used to provide visual feedback on plaque accumulation present and focused tooth brushing advice will be provided at three appointments.

SECONDARY OUTCOMES:
To find difference in demineralisation (ΔF) between the White light group and QLF groups from visit 1 to visit 3. | 6 Months
  The difference in demineralisation (ΔF) between the White light group and QLF groups from visit 1 to visit 3 will be measured. The QLFD camera will take QLF(blue light) and WL (white light) photographs. Either white light image or QLF image (based on which group patient is randomized to will be used to provide visual feedback on the demineralisation present and focused tooth brushing advice will be provided at three appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Norah Flannigan, Principal Investigator — University of Liverpool
Locations (1):
- Dr Norah Flannigan, Liverpool, Merseyside, United Kingdom